CLINICAL TRIAL: NCT02215382
Title: Intraocular Pressure Changes Associated With Tracheal Extubation: Comparison of Sugammadex With Conventional Reversal of Neuromuscular Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, özgür yağan, MD, assistant professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Odu-3
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-08

CONDITIONS: Intraocular Pressure Changes During Tracheal Extubation
Keywords: two reversal methods; changes in IOP; heart rate; blood pressure; tracheal extubation
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- sugammadex (Active Comparator)
  Interventions: Drug: sugammadex
- neostigmine + atropine (Active Comparator)
  Interventions: Drug: neostigmine+atropine

INTERVENTIONS:
Drug: sugammadex — sugammadex 2 mg/kg
  Arms: sugammadex
Drug: neostigmine+atropine — neostigmine 0,05 mg/kg + atropine 0,025 mg/kg
  Arms: neostigmine + atropine

SUMMARY:
The aim of this study, comparison of effects of sugammadex versus neostigmine/atropine combination on hemodynamic parameters and intraocular pressure during tracheal extubation.

This prospective, randomised study was designed to compare two reversal methods with respect to changes in IOP, heart rate and blood pressure during tracheal extubation period.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status
* elective surgery
* endotracheal intubation under general anesthesia

Exclusion Criteria:

* emergency surgery
* pregnancy
* laparoscopic surgery
* prone position
* BMI > 30 kg/m2
* sedative drug use in last month
* patients with glaucoma.
* ASA > II physical status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | baseline, before applying reversal agent, after applying reversal agent, one, three, five and ten minutes after tracheal extubation

SECONDARY OUTCOMES:
heart rate | baseline, before applying reversal agent, after applying reversal agent, one, three, five and ten minutes after tracheal extubation
blood pressure | baseline, before applying reversal agent, after applying reversal agent, one, three, five and ten minutes after tracheal extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Reanimation Dept. Ordu University Training and Research Hospital, Altinordu, Ordu, Turkey (Türkiye)